CLINICAL TRIAL: NCT01960530
Title: An Open Label, Partially Randomised, Single Dose, Crossover Study to Evaluate the PK, Oral Bioavailability and Relationship to Metabolic Parameters of Hydrocortisone and Infacort® in Healthy Adult Male Volunteers.
Brief Title: An Investigational Study of Hydrocortisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Infacort 002
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Endogenous Cortisol (No Intervention): No Study medication will be given during this study period, however various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
- Dexamethasone (Other): 1mg Dexamethasone will be administered at 22:00 on Day 1 and at 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points. Dexamethasone is considered a challenge agent and therefore a non-IMP
  Interventions: Other: Dexamethasone
- Infacort® (Experimental): 20mg Infacort® will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous adrenocorticotropic Hormone (ACTH) and cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Interventions: Drug: Hydrocortisone granules
- Hydrocortisone Tablet (Active Comparator): 20mg Hydrocortisone Tablet will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous ACTH and Cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Interventions: Drug: Hydrocortisone Tablet
- i.v Hydrocortisone Injection (Active Comparator): 20mg i.v. Hydrocortisone Injection will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous ACTH and Cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Interventions: Drug: i.v. Hydrocortisone Injection

INTERVENTIONS:
Drug: Hydrocortisone granules — Multi-particulate granules
  Other Names: Infacort
  Arms: Infacort®
Drug: Hydrocortisone Tablet — Standard hydrocortisone tablets
  Other Names: Commerical supply
  Arms: Hydrocortisone Tablet
Drug: i.v. Hydrocortisone Injection — Standard hydrocortisone solution for intravenous injection
  Other Names: Commerical supply
  Arms: i.v Hydrocortisone Injection
Other: Dexamethasone — Challenge agent
  Other Names: Non-IMP
  Arms: Dexamethasone

SUMMARY:
This study will investigate a new drug called Infacort®; a newly-developed immediate release formulation of a well-established drug called hydrocortisone. Hydrocortisone is used as a replacement treatment for people whose adrenal glands are not producing enough natural cortisol - a condition known as adrenal insufficiency. The study will assess how Infacort® acts once inside the body, by measuring cortisol and other hormone levels in the body, compared to already marketed hydrocortisone tablet and hydrocortisone intravenous (through the vein) injection.

The population who are eligible to take part in the study are healthy male volunteers, aged between 18 and 60 years of age.

DETAILED DESCRIPTION:
The study will evaluate the normal physiology, PK and metabolism of cortisol, investigate the PK and bioavailability of cortisol from the test Infacort® Granules (hydrocortisone) and the reference hydrocortisone tablets and i.v injection in healthy adult male volunteers and explore the role of cortisol in the regulation of metabolic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 60 years of age, inclusive (at screening).
* Subjects with a Body Mass Index (BMI) of 21-28. Body Mass Index = Body weight (kg) / (Height (m))*2.
* Subjects with no clinically significant abnormal serum biochemistry, haematology and urinalysis values within 14 days prior to Day 1 of Study Period 1.
* Subjects with a negative urinary drugs of abuse screen, determined within 14 days prior to Day 1 of Study Period 1. A positive alcohol test may be repeated at the discretion of the Investigator.
* Subjects with negative HIV and Hepatitis B and C results.
* Subjects with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 14 days prior to Day 1 of Study Period 1.
* Subjects with no clinically-significant deviation outside the normal ranges for blood pressure and pulse measurements.
* Subjects (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) and sexual partners must use effective contraception methods during the trial and for 3 months after the last dose, for example:

  * Oral contraceptive + condom
  * Intra-uterine device (IUD) + condom
  * Diaphragm with spermicide + condom
* Subjects must be available to complete the study.
* Subjects must satisfy a medical examiner about their fitness to participate in the study.
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication within 14 days prior to Day 1 of Study Period 1 (including high dose vitamins, dietary supplements or herbal remedies).
* Receipt of any vaccination within 14 days prior to Day 1 of Study Period 1.
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Presence of clinically significant infections (systemic fungal and viral infections, acute bacterial infections).
* Current or previous history of tuberculosis.
* A clinically significant history of previous allergy / sensitivity to Hydrocortisone and/or Dexamethasone.
* A clinically significant history or family history of psychiatric disorders/illnesses.
* A clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. The washout period between trials is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study)
* Subjects who have consumed more than 2 units of alcohol per day within seven (7) days prior to Day 1 of Study Period 1or have consumed any alcohol within the 48 hour period prior to Day 1 of Study Period 1.
* Donation of 450ml or more of blood within the previous 3 months.
* Subjects who smoke (or ex-smokers who have smoked within 6 months prior to Day 1 of Study Period 1).
* Subjects who work shifts (i.e. regularly alternate between days, afternoons and nights).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-period Crossover: Study Period 1 (Endogenous Cortisol): No IMP was administered. Subjects were observed over a 24 hour period, during which sleep disruption was minimised, to record their endogenous cortisol production as a baseline figure and to confirm eligibility for the subsequent study periods.
  Study Period 2 (Dexamethasone): Subjects were admitted to the unit following a final confirmation of eligibility, prior to administration with Dexamethasone.
  Study Periods 3 and 4 (Infacort Granules or Hydrocortisone Tablets): Subjects were admitted to the unit and ongoing eligibility was confirmed. Subjects received both treatments (1 in Period 3, and 1 in Period 4), and were randomised using the PROC PLAN procedure of SAS. Subjects received Dexamethasone 1 hour prior to IMP administration.
  Study Period 5 (I.V. Hydrocortisone Injection): Subjects were admitted to the unit and ongoing eligibility was confirmed. Subjects received Dexamethasone 1 hour prior to IMP administration.
Period: Overall Study
Arm/Group | 5-period Crossover
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- All Participants: All participants received no IMP, dexamethasone (non-IMP), oral infacort, oral hydrocortisone, i.v. hydrocortisone
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: Derived PK for Serum Cortisol: Maximum serum concentration (Cmax)
Time Frame: Hourly from 0 to 24 hours
Population: All randomised subjects who received no IMP (no treatment), dexamethasone, oral Infacort®, hydrocortisone tablet and i.v. hydrocortisone, had sufficient serum cortisol concentration by time profiles and who did not violate the protocol
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Groups:
- Infacort®: 20mg Infacort® will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous Adrenocorticotropic Hormone(ACTH)and Cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Infacort
- Hydrocortisone Tablet: 20mg Hydrocortisone Tablet will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous ACTH and Cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Hydrocortisone Tablet
- i.v Hydrocortisone Injection: 20mg i.v. Hydrocortisone Injection will be administered on Day 2 at 07:00. Dexamethasone is a challenge agent and will be taken to suppress endogenous ACTH and Cortisol. 1mg Dexamethasone will be administered at 22:00 on Day 1 and 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  i.v. Hydrocortisone Injection
Arm/Group | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 14 | 14
nmol/L | 940.012 (283.773) | 896.489 (258.083) | 1563.479 (491.267)
Statistical Analysis 1: Comparison: Infacort® vs i.v Hydrocortisone Injection; Evaluation of Cmax; Test type: Non-Inferiority or Equivalence — To investigate the absolute and relative bioavailability of cortisol from oral Infacort®, a 20 mg dose of oral Infacort® was compared to a 20 mg dose of i.v. hydrocortisone and hydrocortisone tablets, respectively (Study Periods 3-5). These investigations were conducted in dexamethasone suppressed healthy subjects. Standard bioavailability limits of 80% to 125% were used; Geometric LSmean ratio = 60.12, 90% CI 2-sided [54.69 to 66.10]
Statistical Analysis 2: Comparison: Infacort® vs Hydrocortisone Tablet; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LSmean ratio = 106.83, 90% CI 2-sided [96.92 to 117.76]

2. Secondary Outcome: Adverse Events (AEs)
Description: Number of subjects with adverse events throughout the study.
Time Frame: Days 1-2 during each Study Period
Measure: Number; unit: participants
Groups:
- Dexamethasone: 1mg Dexamethasone will be administered at 22:00 on Day 1 and at 06:00 and 12:00 on Day 2. Various blood, urine and saliva samples will be taken in order to measure normal levels of hormones and other chemicals at several time-points.
  Dexamethasone
Arm/Group | Endogenous Cortisol | Dexamethasone | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
participants | 3 | 3 | 0 | 1 | 2

3. Secondary Outcome: Concentrations of Cortisol Binding Protein
Description: Cortisol protein binding under physiological conditions and after the administration of dexamethasone and hydrocortisone.
Time Frame: Blood samples on Day 1 and/or Day 2 of each Study Period
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Endogenous Cortisol | Dexamethasone | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
ug/mL | 22.950 (2.7355) | 23.441 (3.0381) | 22.386 (2.8753) | 21.757 (3.6545) | 21.482 (3.2047)

4. Secondary Outcome: Insulin Sensitivity Under Physiological Conditions and After Administration of Dexamethasone and Infacort®, Hydrocortisone Tablets and i.v Hydrocortisone.
Description: A standardised mixed meal elevates blood glucose and provides a reproducible stimulation of insulin release. Lower levels of insulin secretion, whilst maintaining normoglycaemia would indicate enhanced insulin sensitivity and glucose disposal; higher insulin levels will reflect insulin resistance.
Time Frame: Blood samples on Day 1 and/or Day 2 of each Study Period
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Endogenous Cortisol | Dexamethasone | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
uIU/mL | 70.529 (17.975) | 80.668 (40.801) | 77.575 (32.195) | 70.650 (34.983) | 70.121 (27.140)

5. Secondary Outcome: PK and Metabolism of Cortisol
Description: Blood: Serum cortisol under physiological conditions and after administration of dexamethasone and Infacort® Granules, Hydrocortisone Tablets and i.v Hydrocortisone Injection.
Time Frame: Blood, urine & saliva samples on Day 1 and/or Day 2 of each Study Period
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Endogenous Cortisol | Dexamethasone | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
nmol/L | 447.355 (77.005) | 19.349 (9.567) | 963.134 (283.376) | 893.077 (259.730) | 1580.337 (492.285)

6. Primary Outcome: AUC0-t
Description: Derived PK for Serum Cortisol: Area under the curve from 0-24 hours
Time Frame: Hourly from 0 to 24 hours
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Number analyzed (Participants) | 14 | 13 | 14
nmol*h/L | 2543.24 (713.76) | 2896.73 (850.31) | 2923.46 (971.41)
Statistical Analysis 1: Comparison: Infacort® vs i.v Hydrocortisone Injection; Test type: Superiority or Other; Mean Difference (Final Values) = 86.99, 90% CI 2-sided [79.23 to 95.52]
Statistical Analysis 2: Comparison: Infacort® vs Hydrocortisone Tablet; Test type: Superiority or Other; Mean Difference (Final Values) = 89.96, 90% CI 2-sided [81.72 to 99.04]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Endogenous Cortisol | Dexamethasone | Infacort® | Hydrocortisone Tablet | i.v Hydrocortisone Injection
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 3/14 | 0/14 | 1/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endogenous Cortisol (N=14) | Dexamethasone (N=14) | Infacort® (N=14) | Hydrocortisone Tablet (N=14) | i.v Hydrocortisone Injection (N=14)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must obtain written consent from the Sponsor prior to any publication of results.